CLINICAL TRIAL: NCT05313165
Title: Percutaneous Deep Vein Arterialization for the Treatment of Late-Stage Chronic Limb-Threatening Ischemia: The PROMISE III Trial
Brief Title: PROMISE III: Percutaneous Deep Vein Arterialization for the Treatment of Late-Stage Chronic Limb-Threatening Ischemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LimFlow, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LF-CA-PR-53
Record Dates: First submitted 2022-03-12; First posted 2022-04-06 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Critical Limb Ischemia; Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease
Keywords: CLTI; PAD; CLI
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treated with LimFlow (Experimental): Treatment with the LimFlow Stent Graft System
  Interventions: Device: LimFlow Stent Graft System

INTERVENTIONS:
Device: LimFlow Stent Graft System — Creation of an arteriovenous fistula in the desired limb location

SUMMARY:
A prospective, single-arm, multi-center study designed to gather additional information on the LimFlow System.

DETAILED DESCRIPTION:
The objective of this study is to provide additional information on the LimFlow System for creating an AV connection in the Below The Knee (BTK) vascular system using an endovascular, minimally invasive approach to arterialize the pedal veins for the treatment of chronic limb-threatening ischemia in subjects ineligible for conventional endovascular or surgical limb salvage procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥ 18 and ≤ 95 years of age
2. Clinical diagnosis of chronic limb-threatening ischemia, defined as any of the following clinical assessments: previous angiogram or hemodynamic evidence of severely diminished arterial inflow of the index limb (e.g., ABI ≤ 0.39, TP / TcPO2 < 30 mm Hg) and

   1. Rutherford Classification 5, ischemic ulceration or
   2. Rutherford Classification 6, ischemic gangrene
3. Subject has been assessed by the Principal Investigator and determined that no conventional distal bypass, surgical or endovascular therapy for limb salvage is feasible due to either a) absence of a usable pedal artery target (endovascular or surgical approach), or b) the presence of a pedal artery target with absence of a viable single-segment vein in either lower extremity or either arm that could be used for autogenous vein conduit.
4. Proximally, the Target In-flow Artery at the cross-over point must fall within the recommended vessel diameter ranges for the LimFlow stent graft by visual estimation.
5. Subject is willing and able to sign the informed consent form.
6. Subject is enrolled in an acceptable wound care network and has an adequate support network to ensure that subject is compliant with medication regimen and follow-up study visits.
7. Prior to enrollment (7-day window), women of childbearing potential must have a negative pregnancy test.
8. Primary wound is stable (e.g., not rapidly deteriorating and/or showing signs of healing).
9. Stable glycemic control, HbA1C < 10% (<269mg/dL)
10. Subjects requiring dialysis may be included, provided they meet all the following requirements:

    * On dialysis for > 6 months
    * Autologous arteriovenous (AV) fistula or peritoneal access used for hemodialysis
    * Serum albumin > 30 g/liter
    * BMI > 20

Exclusion Criteria:

1. Concomitant hepatic insufficiency, thrombophlebitis in the target limb, or non-treatable coagulation disorder within the past 90 days.
2. Active immunodeficiency disorder or currently receiving immunosuppressant therapy for an immunodeficiency disorder.
3. Prior peripheral arterial bypass procedure above or below the knee which would inhibit proximal inflow to the stent graft.
4. Absence of adequate viable tissue in target foot.
5. Life expectancy less than 12 months.
6. Documented myocardial infarction or stroke within previous 90 days.
7. Active infection (e.g., fever, significantly elevated WBC count >20.0 x 109/L, and/or positive blood culture) at the time of the index procedure that may preclude insertion of a prosthesis or require major amputation (e.g., osteomyelitis proximal to metatarsals).
8. Known or suspected allergies or contraindications to aspirin or P2Y12 inhibitors, heparin, stainless steel, nitinol or contrast agent that cannot be adequately pre-treated.
9. Subject is currently taking anti-coagulants, which in the opinion of the investigator, interferes with the subject's ability to participate in the study (i.e., intermittent interruption of therapy for procedure may compromise subject's safety).
10. Lower extremity vascular disease that may inhibit the procedure and/or jeopardize wound healing (e.g., vasculitis, Buerger's disease, significant edema in the target limb, deep venous thrombus in the target vein, hyperpigmentation, or medial ulceration above the ankle).
11. Significant acute or chronic kidney disease with a serum creatinine of > 2.5 mg/dl in subjects not undergoing dialysis.
12. Severe heart failure (e.g., NYHA Class IV), which in the opinion of the investigator may compromise subject's ability to safely undergo a percutaneous procedure.
13. Any significant concurrent medical, psychological, or social condition, which may significantly interfere with the subject's optimal participation in the study, in the opinion of the investigator.
14. The subject is currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.
15. Subject is unwilling, unable, or unlikely for cognitive or social reasons to comply with any of the protocol or follow-up requirements.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Amputation Free Survival | 6 Months
  Freedom from major (above-ankle) amputation and death (all-cause mortality)

SECONDARY OUTCOMES:
Primary Patency | 30 Days
  Absence of occlusion of the endovascular intervention that is maintained without the need for additional or secondary surgical or endovascular procedures
Primary Patency | 6 Months
  Absence of occlusion of the endovascular intervention that is maintained without the need for additional or secondary surgical or endovascular procedures
Primary Assisted Patency | 30 Days
  Absence of occlusion of the endovascular intervention maintained with the use of additional or secondary surgical or endovascular procedures, as long as occlusion of the primary treated site has not occurred
Primary Assisted Patency | 6 Months
  Absence of occlusion of the endovascular intervention maintained with the use of additional or secondary surgical or endovascular procedures, as long as occlusion of the primary treated site has not occurred
Secondary Patency | 30 Days
  Absence of occlusion of the endovascular intervention that is maintained with the use of additional or secondary surgical or endovascular procedures after occlusion occurs
Secondary Patency | 6 Months
  Absence of occlusion of the endovascular intervention that is maintained with the use of additional or secondary surgical or endovascular procedures after occlusion occurs
Limb Salvage | 30 Days
  Percentage of subjects with freedom from above-ankle amputation of the index limb
Limb Salvage | 3 Months
  Percentage of subjects with freedom from above-ankle amputation of the index limb
Limb Salvage | 6 Months
  Percentage of subjects with freedom from above-ankle amputation of the index limb
Change in Rutherford Classification | 30 Days
  A change of one class or greater
Change in Rutherford Classification | 3 Months
  A change of one class or greater
Change in Rutherford Classification | 6 Months
  A change of one class or greater
Technical Success | Intraprocedurally
  The successful creation of an arteriovenous fistula in the desired limb location with immediate morphological success
Procedural Success | 30 Days
  The combination of technical success, and absence of all-cause death, above-ankle amputation or clinically driven major re-intervention of the stent graft
Target Wound Healing | 30 Days
  Complete healing of the patient's target wound
Target Wound Healing | 3 Months
  Complete healing of the patient's target wound
Target Wound Healing | 6 Months
  Complete healing of the patient's target wound
Target Wound Healing | 12 Months
  Complete healing of the patient's target wound
All Wound Healing | 30 Days
  Complete healing of the patient's wounds
All Wound Healing | 3 Months
  Complete healing of the patient's wounds
All Wound Healing | 6 Months
  Complete healing of the patient's wounds
All Wound Healing | 12 Months
  Complete healing of the patient's wounds
All Wound Area Reduction | 30 Days
  Reduction in area of the patient's wounds
All Wound Area Reduction | 3 Months
  Reduction in area of the patient's wounds
All Wound Area Reduction | 6 Months
  Reduction in area of the patient's wounds
All Wound Area Reduction | 12 Months
  Reduction in area of the patient's wounds
Freedom from Contrast-Induced Nephropathy | 72 hours
  Subjects without acute (within 72 hours after intravenous contrast administration) impairment of renal function, measured as an absolute ≥0.5 mg/dL (44 μmol/L) increase compared to baseline SCr value that results in a value above the upper limit of the normal range.
Procedure Time | Intraprocedurally
  The time of the first puncture (venous or arterial) to when the last catheter is removed
Radiation Exposure | Intraprocedurally
  Patient radiation exposure (in milligray) during the procedure
Contrast Volume | Intraprocedurally
  The total volume of contrast media (in milliliters) given during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Clair, MD, Principal Investigator — Vanderbilt University; Mehdi Shishehbor, Principal Investigator — University Hospital Cleveland
Locations (30):
- United States (30):
  - University of California, San Diego Health, La Jolla, California
  - Stanford University School of Medicine, Palo Alto, California
  - UCSF, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Yale University, New Haven, Connecticut
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - UMass Chan Medical School, Worcester, Massachusetts
  - Washington University / Barnes Jewish, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Vascular Institute of Atlantic Medical Imaging, Pomona, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Presbyterian Healthcare, Albuquerque, New Mexico
  - Northwell Health Long Island Jewish Medical Center, Lake Success, New York
  - NYU Langone Health, New York, New York
  - Mount Sinai, New York, New York
  - Cornell University, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Penn State Health, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Ascension Columbia St. Mary's Hospital, Milwaukee, Wisconsin
  - The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
No plan to share